CLINICAL TRIAL: NCT03437616
Title: Cardiovascular Rehabilitation - Effectiveness of the Tulppa Program - a Controlled Study
Brief Title: Cardiovascular Rehabilitation - Effectiveness of the Tulppa Program
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rehabilitation Foundation, Finland (Other)
Collaborators: Finnish Heart Association (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tulppa-40310
Record Dates: First submitted 2018-01-10; First posted 2018-02-19 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Coronary Heart Disease
Keywords: Rehabilitation; Coronary heart disease; Cardiovascular diseases; Risk factors; Life-style changes; Efficacy
MeSH Terms: conditions — Coronary Disease; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Longitudinal controlled study: The intervention group (n=150) participates in Tulppa rehabilitation program and the control group (n=150) do not participate in Tulppa rehabilitation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tulppa rehabilitation (Experimental): 8-10 weekly 3-hour group sessions and two follow-up sessions (6 and 12 months).
  Interventions: Behavioral: Tulppa rehabilitation
- Control group (No Intervention): Control group does not receive Tulppa rehabilitation during the study.

INTERVENTIONS:
Behavioral: Tulppa rehabilitation — The intervention includes health education on e.g. healthy diet, weight management, physical activity and psychosocial coping as well as peer discussions and physical exercises.
  Arms: Tulppa rehabilitation

SUMMARY:
This study investigates the effectiveness of a Finnish Tulppa outpatient rehabilitation program. Tulppa is a group-based secondary prevention program for patients with vascular diseases. The program is developed by the Finnish Heart Association. The intervention is implemented at the local primary health care centers in 12 health districts in Finland.

A longitudinal controlled study is used to investigate the effects of the intervention on participants' level of cardiovascular risk factors (e.g. lipids, blood pressure, body mass index), functional capacity (e.g. 6 minute walk test), life style as well as psychosocial factors (e.g. smoking, diet, physical activity, health-related quality of life and depression). The data will be collected at baseline (i.e. before the intervention), and 6 and 12 months after the intervention started.

The participants (n = 300) are patients diagnosed with coronary heart disease. The study group (n = 150) is recruited from participants of Tulppa rehabilitation in three health care districts (Pirkanmaa, South Karelia, Päijät-Häme). The control group (n = 150) is recruited from two health care districts (Turku and Hyvinkää) that do not provide Tulppa rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Study group: Patients diagnosed with coronary heart disease taking part in the Tulppa cardiac rehabilitation program at Pirkanmaa, South Karelia and Päijät-Häme health districts
* Control group: Patients diagnosed with coronary heart disease, living in the area of Turku or Hyvinkää which are health districts that do not provide Tulppa rehabilitation.

Exclusion Criteria:

* Acute and severe mental health problems, alcohol abuse, major limitations in physical activities

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-02-19 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Health related quality of life | Changes between baseline, 6 months and 12 months
  Health related quality of life is assessed with the finnish version of RAND-36-Item Health Survey (36-Item Short Form Survey Instrument - SF-36; Aalto, Aro & Teperi, 1999). The RAND-36 is a generic health-related survey consisting of 36 items with eight sub-scales: 1. general health, 2. bodily pain, 3. physical functioning, 4. role limitations/physical, 5. role limitations/emotional, 6. vitality, 7. mental health, and 8. social functioning. The total score is a sum of the eight subscales and the range is 0 - 100. Higher scores on the scale indicate a better quality of life.
Modified North Karelia CVD risk score | Changes between baseline, 6 months and 12 months
  The limit values to calculate the CVD risk score were originally developed during the North Karelia project (Puska et al., 2009) and were further elaborated by Ketola (2001). The modified CVD risk score consists of six risk factors:
  1. Body mass index (BMI)
  2. Smoking
  3. Physical inactivity
  4. Systolic blood pressure
  5. Diastolic blood pressure
  6. Total cholesterol. The total score of the index is a sum of the 6 risk factors and the range is 0-16, the cut-off point indicating high risk of CVD is 4.5. Higher scores on the scale indicate a higher risk of cardiovascular disease. Subscore outcomes of the CVD risk score are defined as secondary outcome measures below.

SECONDARY OUTCOMES:
The 6-Min Walk Test | Changes between baseline, 6 months and 12 months
  The 6-min Walk Test (6MWT) measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes.
Blood pressure | Changes between baseline, 6 months and 12 months
  Blood pressure is expressed in terms of the systolic and diastolic pressure and is measured in millimeters of mercury (mmHg).
Waist circumference | Changes between baseline, 6 months and 12 months
  Waist circumference is measured halfway between the costal margin and iliac crest in centimeters.
Body mass index | Changes between baseline, 6 months and 12 months
  The body mass index (BMI) is calculated as weight in kilograms divided by height in meters squared (kg/m2).
Lipid profile | Changes between baseline, 6 months and 12 months
  Triglycerides, LDL-, HDL- and total cholesterol level will be measured with laboratory test
Blood glucose level | Changes between baseline, 6 months and 12 months
  Fasting plasma glucose (mmol/l) will be measured with laboratory test
Physical inactivity | Changes between baseline, 6 months and 12 months
  Physical inactivity is assessed with one question about the frequency per week of physical exercise causing swetting and /or some shortness of breath (1 = 3 or more times/week, 2 = 1-2 times/week, 3 = 1 time/week, 4 = sometimes, 5 = never)
Smoking | Changes between baseline, 6 months and 12 months
  Smoking is evaluated with one question about number of cigarettes/day (0 = not at all...8 = 30 or more cigarettes/day)
Alcohol use | Changes between baseline, 6 months and 12 months
  Alcohol use is measured with two questions:
  1. How often do you have drinks containing alcohol? (0 = never, 1 = monthly or less, 2 = 2-4 times a month, 3 = 2-3 times a week, 4 = 4 times a week or more)
  2. How many drinks containing alcohol do you have on a typical day when you are drinking? (1 = 1-2 drinks, 2 = 3-4, 3 = 5-6, 4 = 7-9, 5 = 10 drinks or more)
Dietary habits | Changes between baseline, 6 months and 12 months
  Dietary habits are evaluated with 3 questions:
  Do you eat regular meals? (2 = yes, 1 = I don´t know, 0 = no) Do you use low-fat foods? (2 = yes, 1 = I don´t know, 0 = no) Do you eat enough good / healthy fat? (2 = yes, 1 = I don´t know, 0 = no)
Depression | Changes between baseline, 6 months and 12 months
  Depression will be measured using The finnish Depression Scale DEPS (Salokangas, R. K., Poutanen, O & Stengard, E.,1995). 10 items, the items are rated from 0 to 3 (0 = not at all... ...3 = very much) and the range of the total score is 0-30. Higher scores on the scale indicate a higher probability of depression.
Anxiety | Changes between baseline, 6 months and 12 months
  Anxiety will be assessed with the state-anxiety sub-scale of the Endler Multidimensional Anxiety Scales (EMAS-State) (Endler, N. S., Parker, J. D. A., Bagby, R. M., & Cox, B. J., 1991). The State-anxiety sub-scale consists of 20 items evaluated on a five-point Likert scale (score range 20-100). EMAS-State assesses two components of state-anxiety : a cognitive worry component and an autonomic-emotional component. Both components consist of ten items. In this study the 10 items of a cognitive worry component is used. Higher scores indicate a higher level of cognitive worry.

OTHER OUTCOMES:
Family support | Baseline, 6 months and twelve months
  Partner support will be measured with a Finnish 12-item Family Support (FS) scale (Julkunen & Greenglass, 1989; Gustavsson-Lilius M., Julkunen J., & Hietanen P., 2007). The items are rated using a five-step Likert scale (1 = completely disagree… 5 = completely agree) and the range of the total score is 12 - 60. The sum-score of the scale reflects the respondents' perceived degree of emotional and instrumental support received from other family members. Higher scores on the scale indicates higher amount of perceived support from the family.

CONTACTS AND LOCATIONS:
Overall Officials: Erja Poutianen, PhD, Study Director — Rehabilitation Foundation; Mila Gustavsson-Lilius, PhD, Principal Investigator — Rehabilitation Foundation; Piia Pietilä, MA, Principal Investigator — Rehabilitation Foundation
Locations (1):
- Rehabilitation Foundation, Helsinki, Malminkartano, Finland